CLINICAL TRIAL: NCT00063973
Title: Phase I Study of Cilengitide (EMD 121974) in Children With Refractory Brain Tumors
Brief Title: Cilengitide in Treating Children With Refractory Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03175; NCI-2012-03175 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR653715; PBTC-012 (Other: Pediatric Brain Tumor Consortium); PBTC-012 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Childhood Central Nervous System Germ Cell Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Brain Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma | interventions — Cilengitide

ARMS (1):
- Treatment (cilengitide) (Experimental): Patients receive cilengitide (EMD 121974) IV over 1 hour twice weekly. Treatment repeats every 4 weeks for 13 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of cilengitide until the MTD is determined. The MTD is defined as the dose at which 25% of patients are expected to experience dose-limiting toxicity. Once the MTD is determined, 6 additional patients are accrued and treated at that dose level for a total of 12 patients at the MTD.
  Interventions: Drug: cilengitide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of cilengitide in treating children with recurrent, progressive, or refractory primary CNS tumors. Cilengitide may slow the growth of brain cancer cells by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the acute and dose-limiting toxicities (DLT) and define the maximum tolerated dose (MTD) of cilengitide (EMD 121974) when administered to children and adolescents with refractory primary brain tumors.

SECONDARY OBJECTIVES:

I. To obtain preliminary evidence of biologic activity by determining alterations in tissue perfusion, tumor blood flow and metabolic activity using MR perfusion, PET and MRS and correlating these findings with changes in tumor size by volumetric MRI.

II. To characterize inter- and intra-patient variability in the pharmacokinetics of cilengitide and to estimate cilengitide renal clearance in this patient population.

III. To characterize the pharmacogenetic polymorphisms in drug transporters (e.g., MRP4, BCRP) and relate to cilengitide disposition.

IV. To evaluate changes in circulating endothelial cells (CECs) and circulating endothelial precursors (CEPs) in patients treated with cilengitide, and to investigate the correlation between changes in CECs and CEPs, plasma, serum and urine angiogenic protein levels such as VEGF, and clinical outcome.

V. To obtain preliminary information about the efficacy of cilengitide in this patient population.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive cilengitide (EMD 121974) IV over 1 hour twice weekly. Treatment repeats every 4 weeks for 13 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cilengitide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 25% of patients are expected to experience dose-limiting toxicity. Once the MTD is determined, 6 additional patients are accrued and treated at that dose level for a total of 12 patients at the MTD.

Patients receiving treatment are followed weekly for the first three months then monthly for one year or 13 courses of treatment. Patients discontinuing treatment will be followed for resolution of all adverse events occurring while on treatment and/or within 30 days of the last administration of study drug.

Patients will be followed for the shortest of 1) three months after the last protocol based treatment, or 2) the date other therapy is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of primary CNS tumor and evidence that the tumor is recurrent or progressive and refractory to standard therapy, including histologically benign CNS tumors (e.g. low-grade glioma); clinical and radiographic evidence of a brain stem or optic pathway glioma is required in the absence of histologic diagnosis
* Karnofsky or Modified Lansky Score ≥ 50%
* Patients with neurological deficits should have deficits that are stable for ≥ 1 week prior to study entry
* Chemotherapy: Patients with evidence of recovery from prior therapy; no investigational agent, including biologic agent, within two (2) weeks of study entry; at least six (6) weeks from nitrosourea agent to study entry; at least four (4) weeks from any myelosuppressive therapy to study entry
* Bone Marrow Transplant: Greater than six (6) months prior to study entry
* XRT: At least six (6) weeks from prior radiation therapy to study entry; greater than three (3) months from prior craniospinal irradiation (> 24 Gy) or total body irradiation to study entry; greater than two (2) weeks from local palliative irradiation to study entry
* Anti-convulsants: Patients will be eligible for this study even if they are receiving anti-convulsants
* Growth factors: Off all colony forming growth factor(s) > one (1) week prior to study entry (G-CSF, GM-CSF, erythropoietin)
* Corticosteroids: Patients receiving corticosteroids must be receiving a stable dose for ≥ one (1) week prior to study entry
* ANC > 1,000/μl
* Platelets > 100,000/μl (transfusion independent)
* Hemoglobin > 8.0 g/dl (may be transfused)
* Patients with bone marrow involvement may be eligible
* Creatinine < 1.5 times normal range for age
* GFR > 70 ml/min/1.73m^2
* Total bilirubin ≤ upper limit of normal for age
* SGPT (ALT) and SGOT (AST) < 2.5 times upper limit of normal
* Cilengitide was teratogenic when tested in animals; as such, female patients of childbearing potential must have a negative serum or urine pregnancy test prior to study entry; female patients must avoid breast feeding while on study
* Patients of childbearing potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Signed informed consent according to institutional guidelines must be obtained prior to patient registration

Exclusion Criteria:

* Patient must not be receiving any other anticancer or experimental drug therapy, with the exception of corticosteroids
* Patient must have no uncontrolled infection
* Patient has no overt renal, hepatic, cardiac or pulmonary disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
MTD of cilengitide | 4 weeks

SECONDARY OUTCOMES:
Response | Up to 3 months
  Reported and recorded descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Tobey MacDonald, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States